CLINICAL TRIAL: NCT05079763
Title: Bacterial Cellulose-monolaurin Hydrogel for Preventing Therapy-induced High-grade Acute Dermatitis Among Filipinos With Breast Adenocarcinoma: a Pilot Randomized Controlled Trial
Brief Title: Bacterial Cellulose-monolaurin Hydrogel for Acute Radiation Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UPMREB 2021-140-01
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Radiation Dermatitis
Keywords: ARD; postmastectomy; breast cancer; breast adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Bacterial cellulose-monolaurin hydrogel
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Application of bacterial cellulose-monolaurin hydrogel in the prescribed area for every 12 hours starting from receipt of first radiotherapy until development of moist desquamation or two week after completion of radiotherapy plan
  Interventions: Other: Bacterial cellulose-monolaurin hydrogel
- Placebo Arm (Placebo Comparator): Application of placebo cream in the prescribed area for every 12 hours starting from receipt of first radiotherapy until development of moist desquamation or two week after completion of radiotherapy plan
  Interventions: Other: Placebo cream

INTERVENTIONS:
Other: Bacterial cellulose-monolaurin hydrogel — Hydrogel containing Komagataeibacter xylinus-derived bacterial cellulose, virgin coconut oil monolaurin, cucumber fragrance and distilled water
  Arms: Experimental arm
Other: Placebo cream — Cream containing distilled water, white petrolatum, steady alcohol, propylene glycol, sodium laurel sulphate, methylparaben and propylparaben
  Arms: Placebo Arm

SUMMARY:
Acute radiation dermatitis (ARD) is almost universally experienced by patients with cancer during or after radiation therapy. This condition potentially leads to detrimental clinical outcomes as it adversely affects adherence to prescribed subsequent management and further worsens quality of life. Nevertheless, there remains no consensus on the appropriate intervention for ARD. This pilot two parallel-group randomized trial aims to clinically assess the potential of bacterial cellulose-monolaurin hydrogel, compared to placebo cream, to prevent high-grade ARD among Filipinos with breast cancer up to four weeks after last radiotherapy session.

ELIGIBILITY:
Inclusion Criteria:

* Female sex at birth
* Age at least 18 years at the time of invitation
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of either 0 or 1
* With histopathologic diagnosis of breast carcinoma
* Already completed prescribed mastectomy and chemotherapy (adjuvant or neoadjuvant) interventions
* Scheduled to receive hypo fractionated postmastectomy-postchemotherapy radiation therapy

Exclusion Criteria:

* Pregnant or lactating
* With concurrent or previous history of any malignancy
* With history of mediastinal or thoracic irradiation
* With current bilateral synchronous breast carcinoma
* With diagnosis of metastases from any form of breast cancer
* With any skin lesion in the planned radiation field deemed deramtologically and/or radiotherapeutically relevant
* With concomitant disease states deemed clinically significant (connective tissue diseases, infections, uncontrolled chronic disorders, renal failure, hepatic dysfunction, etc.)
* With known history of hypersensitivities and/or reactions against any component of either experimental or comparator interventions
* Inability to personally provide informed consent or to personally comply with skin care instructions

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of high grade acute radiation dermatitis | Baseline to Week 4 post-radiotherapy
  High-grade acute radiation dermatitis is defined as Common Terminology Criteria for Adverse Events (CTCAE) grade of at least 3

SECONDARY OUTCOMES:
Distribution of participants in terms of ARD CTCAE grades | Baseline to Week 4 post-radiotherapy
  Distribution of participants across the ARD CTCAE grades (0-5) in the two interventions will be compared
Patient-reported quality of life | Baseline to Week 4 post-radiotherapy
  Outcome will be assessed using the Skindex-16 (SD-16) questionnaire, administered on a weekly basis from baseline up to two weeks post-radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Philippine General Hospital, Manila, Philippines